CLINICAL TRIAL: NCT07088770
Title: TechMPower: Advancing HIV/SUD Care and Service Delivery for People Involved in the Criminal Legal System
Brief Title: TechMPower: Advancing HIV/SUD Care and Service Delivery for People in Re-entry
Acronym: TMP Project
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Timothy Hunt, Associate Research Scientist in the Faculty of Social Work, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: AAAV1468; 1R61DA060620-01 (NIH)
Record Dates: First submitted 2025-07-19; First posted 2025-07-28 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: HIV (Human Immunodeficiency Virus); Substance Abuse Disorder
Keywords: People incarcerated in re-entry; HIV testing; Screening, brief intervention, and referral to treatment; Implementation strategies; Implementation team with champion; Navigation case management; Coalition; Techmediated
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: TechMPower, informed by PRISM1/RE-AIM implementation science framework, is an intervention that bundles implementation strategies for correctional settings designed to increase delivery of evidence-based practices (EBPs) to prevent adverse HIV-related (new infections, untreated HIV) and SUD-related outcomes (fatal and non-fatal overdose) among individuals detained in jails and reentering the community. The selected EBPs act to increase: 1) HIV screening via universal rapid point-of-care ( POC) testing (policy/practice change in some jail settings) and self-testing education (WHO universal testing/self-testing; 2) Substance Use Disorder (SUD) screening (via universal SBIRT); and 3) linkage to HIV and SUD care/prevention services supported by Navigation Enhanced Case Management (NCM) using hybrid communication (telehealth/tele-harm reduction, video-conference, face-to-face, text/SMS, etc.) approaches.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TechMPower Implementation Strategies (Experimental): TechMPower applies evidence-based Implementation Strategies, including:
  A) data-driven, Community Coalitions and criminal legal system (CLS) focused workgroup informed by the HEALing Communities Study (HCS) Communities That HEAL(CTH intervention); B) Implementation Team led by champions; C) training on optimal person-centered service delivery for service providers/organizations; and D) tech-mediated service delivery, technical assistance, and training to increase: 1) HIV screening/testing via self-testing; 2) SUD screening, brief interview and referral to treatment (SBIRT); and 3) access to and uptake of biomedical HIV and SUD prevention and treatment (PrEP/PEP/ART); overdose education/naloxone distribution [OEND], opioid use disorder medication [MOUD]) delivered through 4) hybrid linkage (telehealth, face-to-face) to services via Navigation Enhanced Case Management (NCM).
  Interventions: Behavioral: Community Coalition CLS Workgroup/Network of Providers; Behavioral: Tech-mediated Training and Service Delivery; Behavioral: Multidisciplinary Implementation Team with Champion; Behavioral: Tech-mediated Peer Navigation Enhanced Case management (NCM)

INTERVENTIONS:
Behavioral: Community Coalition CLS Workgroup/Network of Providers — Community Coalition/Network of Providers TechMPower forms the foundation of community engagement in this approach, with membership including PLWH and SUD, sheriffs, within-jail staff, community service providers or other partners who are able to advance the adoption of EBPs within jail and service settings. All coalitions are trained and prepared to drive a planning process at the local level for efficient identification and allocation of resources needed to link people from CLS to a network of community providers for HIV and SUD care and retention. Community coalitions integrate evidence-based (ERIC) strategies: Build coalition; Promote network weaving; Identify/train champions; Conduct consensus discussions that support needed services.
Behavioral: Tech-mediated Training and Service Delivery — Researchers will train all staff, healthcare providers and peer navigators to recognize and reduce stigma in CLS and healthcare settings using a training program informed by MPI Frye and colleagues in the CHHANGE (MH102182-01) intervention, which developed an anti-intersectional stigma training program for CBOs and offers comprehensive training to healthcare and social service organizations. Additionally, researchers will train staff and support protocol enhancements as needed to utilize tech mediated service delivery for NCM in-reach and services coordination in the community. These integrate 5 evidence-based (ERIC) implementation strategies: promote consultation; provide clinical/technical supervision; centralize technical assistance; change physical structure and equipment.
Behavioral: Multidisciplinary Implementation Team with Champion — The multidisciplinary Implementation Team will be comprised of a correctional health nurse, social worker and discharge planner or counselor and corrections officer from the jail. A representative from the community coalition and peer and case manager from NCM will join the team using a tech-mediated platform for conducting the training and for on-going weekly case conferencing addressing system and client level barriers and service planning. The role of the champion from the correctional setting will be to convene meetings focused on fidelity to the intervention components, engagement in shared problem-solving and mediation of administrative issues that may inhibit effective implementation of TechMPower. The champion and implementation team may request technical assistance (TA) or implementation facilitation at any point during implementation. This TA may be provided by the investigative team or outside providers from federal programs.
Behavioral: Tech-mediated Peer Navigation Enhanced Case management (NCM) — Navigation-Enhanced Case Management (NCM) uses Project START, a CDC best evidence intervention as its HIV risk reduction framework. Prior to release, a case manager and peer navigator via telehealth and in-person provide discharge planning and patient education and serves as a liaison to the courts. After release, patient navigators facilitate reentry into community care and provide referrals to HIV medical and SUD care as appropriate (e.g., ART, PrEP, MOUD) and assistance with food, housing, transportation, employment, substance dependence, mental health treatment, and legal issues. TechMPower planned to enhance tracking of linkage during NCM services by integrating reporting along with a web-based platform that tracks assignment of providers and peers and follows for 6 months to capture PRISM linkage and retention in MOUD, HIV and ancillary care.

SUMMARY:
The goal of this clinical study in one NY county is to pilot and refine implementation strategies aimed at improving delivery and uptake of evidence-based practices (EBPs) for HIV prevention/treatment and substance use disorder (SUD) care among incarcerated individuals approaching release with or at risk for HIV and SUD.

The main questions it aims to answer are:

1. How feasible and acceptable are the TechMPower implementation strategies (community coalition workgroups, multidisciplinary implementation team with champion, and tech-mediated training/service delivery with peer navigation) in real-world carceral and reentry settings?
2. To what extent do these strategies improve delivery and uptake of HIV testing with self-testing (HST), pre-exposure prophylaxis (PrEP)/antiretroviral treatment (ART), medications for opioids use disorder (MOUD), and overdose education and naloxone distribution (OEND)?
3. What are the preliminary cost estimates for the implementation strategies and EBPs to inform the larger trial to follow in NY and NJ?
4. What are the preliminary impacts on individual-level outcomes such as HIV testing, linkage to care, and SUD treatment initiation?

Our specific aims for the Phase I protocol presented here is conducted in one county (Ulster County) with a sample (n=50) of detained (prisoners) in their county jail are presented here:

* R61 | Aim 1: Evaluate \ preliminary effectiveness of TechMPower, using mixed methods and a pre-/post-evaluation design, on increasing reach of the EBPs resulting in the following outcomes: (1) SUD and HIV screenings (pre-/post-release); and (2) linkage to SUD prevention/care (MOUD, OEND); and (3) linkage to HIV prevention/care (applying a status-neutral approach) with community service providers post-release. (Effectiveness).
* R61 | Aim 2: Identify how adoption/feasibility, implementation/fidelity and sustainability/maintenance of TechMPower may impact effectiveness of TechMPower outcomes as described in Aim 1 in one (Ulster County) jail using surveys of Implementation Team, jail staff and other key stakeholders. (Implementation)
* R61 | Aim 3: Use implementation mapping to adapt implementation strategies for R33 phase. (Implementation)

DETAILED DESCRIPTION:
HIV prevalence in correctional facilities in the US is about five times greater than in the general population and about 14% of people living with HIV (PLWH) experience incarceration/release every year and 15% of those incarcerated do not know their HIV status. Over 50,000 people are incarcerated in New York state and 1-2% are estimated to be PLWH. Similarly, substance use disorder (SUD) is highly prevalent among criminal-legal system (CLS)-involved people, with an estimated 70-80% of US jail detainees having a SUD are at high risk of relapse, overdose-related mortality and HIV infection post-release. Intervening during incarceration provides an opportunity to address HIV care in hard-to-reach individuals, though more robust interventions and staff training is needed to improve care continuity. Increasing point-of-care rapid testing would maximize HIV detection and results receipt among people in jails, and prepare them with needed knowledge and skills post-release.

To fill this gap, the investigators propose a Regional Research Hub (RRH) and 2-phase, Hybrid Type II effectiveness/implementation study to evaluate the effectiveness of TechMPower, an intervention that bundles implementation strategies to increase delivery of evidence-based intervention (EBPs) to prevent adverse HIV-related (new infection, untreated HIV) and SUD-related outcomes (fatal and non-fatal overdose) among a sample of individuals (n=1200) in 6 New York and New Jersey State County jails. In the first phase submitted in this IRB protocol, the researchers will pilot TechMPower to prepare for the phase two full R33 trial, informed by PRISM/RE-AIM and the health equity framework, by recruiting in one NYS county jail (n=50) and an existing HEALing Communities Study coalition workgroup to evaluate the training on and implementation of the selected EBPs required as standard of care in jails. This record contains the R61 pilot portion.

Researchers will compare outcomes before and after implementation of the strategy bundle to see if TechMPower improves reach, adoption, implementation fidelity, and sustainability of integrated HIV/SUD services.

Participants incarcerated (N=50) will:

1. Complete baseline and 3-month follow-up surveys on HIV/SUD behaviors and care engagement
2. Participate in up to 60-minute qualitative interviews (subset N=8)
3. Receive potential HIV/STI testing, referrals to prevention/treatment, and linkage services including peer navigation enhanced case management (NCM)
4. Receive HIV self-test kit and Naloxone upon release

Stakeholder participants (N=20) will:

1. Complete baseline and 3-month follow-up surveys on HIV/SUD behaviors and care engagement
2. Participate in up to 60-minute qualitative interviews (subset N=8)
3. Receive training in HIV and SUD screening and treatment referral (SBIRT), HST and OEND, person-centered approach to care linkage; tech-mediated training and service delivery; and in NCM
4. Participate in coalition workgroup, implementation team and implementation of NCM

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* speaks and understands English
* report using any illicit drug, in the six months prior to incarceration
* report having had condomless receptive and/or insertive vaginal and/or anal sex without either condom use, AND/OR report another HIV risk in the six months prior to incarceration (i.e. shared syringes, STI+)D
* likely to be released in the next 1-3 months

Exclusion Criteria:

* evidence of significant psychiatric or cognitive impairment that would limit effective participation as confirmed during informed consent assessed during informed consent or confirmed by the MacArthur Competence Assessment Tool
* not fluent in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2024-11-22 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of people incarcerated who have received an HIV test | Baseline and 3 months follow-up
  This is to measure HIV testing (including self-testing) at jail. The number of participants that report in survey at least 1 testing will be tallied. Aggregate reporting on testing from facility will be captured for triangulation.
Number of people detained screened for SBIRT | Baseline and 3 months follow-up
  This is to measure the feasibility, efficacy of Screening, Brief Intervention and Referral to treatment (SBIRT) for SUD at jail. The number of participants that report in survey receiving SBIRT will be tallied. Aggregate reporting on SBIRT from facility will be captured for triangulation.
HIV care access & utilization/ART Use/adherence/viral load/CD4 count | 3-month following pos test result, pre- post release
  Service Use Measure: at least one visit to HIV-focused medical at clinic post release. The number of participants that report in surveys receiving HIV treatment will be tallied. Aggregate reporting on HIV treatment from facility referrals will be captured for triangulation.
Average PrEP oral daily/injectable/episodic PrEP captured in records/chart review; ACASI self-report | Baseline and 3 months follow-up
  This is to measure PrEP use, adherence & discontinuation
PEP uptake rate | Baseline and 3 months follow-up
  This is to measure PEP use by seeing the uptake: starter pack & full treatment provision/fulfillment and adherence, PEP to PrEP transition

SECONDARY OUTCOMES:
Number of clients referred and assessed for NCM | Baseline and 6 months
  This is to measure the feasibility of Navigation Enhanced Case Management (NCM). The number of participants that report in survey receiving NCM will be tallied. Aggregate reporting on NCM service delivery will be captured for triangulation.
Number of people incarcerated receiving OEND | Baseline and 3 months follow-up
  This is to measure the Overdose education and Naloxone Distribution (OEND) feasibility at jail. The number of participants that report in survey receiving OEND will be tallied. Aggregate reporting on OEND service delivery from facility will be captured for triangulation.
Number of staff receiving training on TechMPower integrated SUD/HIV service delivery | Baseline and 6 months follow up
  This is to measure the feasibility of TechMPower techmediated training and HIV/SUD integrated service delivery. This is reported on surveys and aggregate reporting on techmediated training attendance logs for triangulation.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy L Hunt, MSW, PhD, Principal Investigator — Columbia University; Victoria A Frye, MPH, DrPH, Principal Investigator — Columbia University; Nabila El-Bassel, PhD, Principal Investigator — Columbia University
Locations (1):
- Ulster County Jail, Kingston, New York, United States

IPD SHARING:
Plan to Share IPD: No
Protecting data from people incarcerated (prisoners) is of the utmost importance.

REFERENCES:
- See also: NIDA funded four major multisite initiatives to address the myriad issues at the intersection of the criminal justice system and substance use and misuse. These initiatives include: Collaborative Network to End the HIV Epidemic and Address Addiction — https://nida.nih.gov/research/nida-research-programs-activities/justice-system-research
- Available data/document: Study Informational Website — https://sig.columbia.edu/research-projects/techmpower — The Social Intervention Group (SIG), Columbia School of Social Work organizational website announcing the TechMPower study.